CLINICAL TRIAL: NCT07020312
Title: Brain-Computer Interface Visualization Training to Optimize Muscle Activation Following Orthopaedic Surgery: A Blinded Randomized Controlled Trial
Brief Title: Brain-Computer Interface Visualization Training to Optimize Muscle Activation Following Orthopaedic Surgery
Acronym: iBrainTechRCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24021101
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Total Hip Arthroplasty (THA); Total Knee Arthroplasty; Hip Arthroscopy
Keywords: ACLR; THA; TKA; Hip Arthroscopy; Arthrogenic muscle inhibition; Electroencephalography; Gait; Motion Analysis; Biomechanics; Strength
MeSH Terms: interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: The study will have two arms - a 1:1 allocation ratio for the control group and for the intervention group- stratified into four orthopedic surgeries:
  * Anterior Cruciate Ligament Reconstruction (ACLR)
  * Total Knee Arthroplasty (TKA)
  * Total Hip Arthroplasty (THA)
  * Hip Arthroscopy (HA) for Femoroacetabular Impingement Syndrome (FAIS) There will be 30 participants per cohort arm for each procedure, totaling 240 participants for the project.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and physicians will be blinded to group allocation to minimize bias in clinical decision-making and post-operative care. Patients will not be blinded due to the nature of the neurofeedback intervention, which cannot be masked. Both study groups will receive standard rehabilitation, with the only difference being the addition of NFVT in the intervention arm. The neurofeedback sessions will take place within the physical therapy clinic, immediately prior to scheduled physical therapy appointments.
  The team delivering the neurofeedback intervention will be the only personnel aware of group allocation. Treating physicians, physical therapists, outcome assessors, and the statistical analysis team will remain blinded to participant allocation throughout the trial. Statistical analyses will be performed by the Rush Statistical Analysis team, an independent third-party ancillary resource, using a coded dataset to ensure blinding is maintained during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (8):
- Anterior cruciate ligament reconstruction (ACLR) - Experimental (Experimental): Intervention Group: Standard post-surgical rehabilitation therapy + iBrainTech neurofeedback training
  Interventions: Other: Visualization training with neurofeedback; Other: Standard post-surgical rehabilitation therapy
- Anterior cruciate ligament reconstruction (ACLR) - Control (Active Comparator): Control group: Standard post-surgical rehabilitation therapy
  Interventions: Other: Standard post-surgical rehabilitation therapy
- Total knee arthroplasty (TKA) - Experimental (Experimental): Intervention Group: Standard post-surgical rehabilitation therapy + iBrainTech neurofeedback training
  Interventions: Other: Visualization training with neurofeedback; Other: Standard post-surgical rehabilitation therapy
- Total knee arthroplasty (TKA) - Control (Active Comparator): Control group: Standard post-surgical rehabilitation therapy
  Interventions: Other: Standard post-surgical rehabilitation therapy
- Total hip arthroplasty (THA) - Experimental (Experimental): Intervention Group: Standard post-surgical rehabilitation therapy + iBrainTech neurofeedback training
  Interventions: Other: Visualization training with neurofeedback; Other: Standard post-surgical rehabilitation therapy
- Total hip arthroplasty (THA) - Control (Active Comparator): Control group: Standard post-surgical rehabilitation therapy
  Interventions: Other: Standard post-surgical rehabilitation therapy
- Hip arthroscopy (HA) - Experimental (Experimental): Intervention Group: Standard post-surgical rehabilitation therapy + iBrainTech neurofeedback training
  Interventions: Other: Visualization training with neurofeedback; Other: Standard post-surgical rehabilitation therapy
- Hip arthroscopy (HA) - Control (Active Comparator): Control group: Standard post-surgical rehabilitation therapy
  Interventions: Other: Standard post-surgical rehabilitation therapy

INTERVENTIONS:
Other: Visualization training with neurofeedback — This technology uses electroencephalography (EEG) to measure brain activity through passive sensors placed on a cap aligned with the motor and frontal cortices. These sensors detect changes in electrical signals when patients imagine performing rehabilitation movements. The EEG data is sent to a computer, where iBrainTech™ software translates it into a virtual avatar that mimics the imagined actions. This real-time feedback-called neurofeedback-helps patients see how well they are engaging their brain during visualization. By turning the process into a video game controlled by brain signals, the platform motivates patients to focus deeply on visualizing the exercises. Repeated activation of these brain regions may help rebuild neuromuscular pathways, improve muscle control, and reduce the effects of Arthrogenic Muscle Inhibition (AMI), a common issue after orthopedic surgery.
  Arms: Anterior cruciate ligament reconstruction (ACLR) - Experimental; Hip arthroscopy (HA) - Experimental; Total hip arthroplasty (THA) - Experimental; Total knee arthroplasty (TKA) - Experimental
Other: Standard post-surgical rehabilitation therapy — Patients will follow a standard physical therapy protocol. The protocol will be assigned by their respective surgeon who conducted the procedure and will be specific to the procedure that the patient underwent.

SUMMARY:
After orthopedic surgeries like knee or hip replacement, some patients struggle to fully activate their muscles due to a condition called Arthrogenic Muscle Inhibition (AMI). AMI can slow recovery and make physical therapy less effective. This clinical trial is testing whether a special type of brain training-called neurofeedback visualization training-can help improve muscle activation and speed up recovery.

In this study, patients will receive standard physical therapy after surgery. Half of them will also use a device that helps them "visualize" exercises while wearing a cap that reads brain signals (EEG). The cap tracks brain activity when patients imagine doing specific movements. A computer then shows a virtual avatar performing the movements, giving feedback in real time-like a video game controlled by the brain.

The study includes patients recovering from one of four surgeries:

1. Anterior cruciate ligament reconstruction (ACLR)
2. Total knee arthroplasty (TKA)
3. Total hip arthroplasty (THA)
4. Hip arthroscopy (HA) for femoroacetabular impingement (FAI)

The goal is to see if this training improves muscle strength, movement, and daily function more than standard therapy alone. The study will take place at Rush University Medical Center in Chicago and enroll 240 adults, with 60 patients per type of surgery. Each participant will be followed for up to 6 months after surgery and complete strength tests, movement assessments, and questionnaires about their recovery.

The hope is that combining brain training with physical therapy will lead to faster, more complete recoveries and improve how patients move after surgery.

DETAILED DESCRIPTION:
1. Introduction

   Background

   Patients recovering from orthopedic surgical procedures require a comprehensive physical rehabilitation process to help recover pre-operative functional mobility and strength.

   A limiting factor in physical rehabilitation is a patient's inability to activate the involved muscle groups postoperatively, a phenomenon termed Arthrogenic Muscle Inhibition (AMI) [1, 2]. AMI is a complex neurological process where the injury or surgery disrupts sensory and motor neurological pathways, resulting in decreased muscle activation and strength. AMI can be a major obstacle to a patient's return to normal mobility and muscular function [2]. For example, patients who have undergone anterior cruciate ligament reconstruction (ACLR), may experience ineffective quadriceps activation and persistent hamstring contracture, leading to loss of passive and active range of motion (ROM). Even with standard physical therapy rehabilitation, patients with AMI have ineffective recovery due to decreased muscular activation and movement dysfunction [3].

   Visualization training with neurofeedback therapy (NFVT) is a non-invasive method that could be used with standard post-operative physical rehabilitation to decrease AMI and help patients recover pre-operative functional mobility and strength.

   The motor regions of the brain (motor cortex) play a crucial role in planning, controlling, and executing voluntary movements. The motor cortex is not only active during actual movement; mentally rehearsing motor acts without physically moving also activates the motor cortex [4]. For example, one could imagine themselves performing squats without squatting (visualization), this process activates the brain regions related to squatting. Such visualization training can enhance the brain's ability to plan, control and execute movement without physical load on the body [5]. Theoretically, this training could help restore disrupted neurological pathways, leading to reduced AMI and improved patient recovery after surgery [6].

   When a brain region has heightened activity, passive sensors on the scalp can detect the increased electrical activity, this technique is known as electroencephalography (EEG). A computer can process the EEG signal and provide users with real time feedback on their concentration level and whether they are activating their motor cortex through mental visualization of movements (neurofeedback). This feedback process enhances the visualization training [6].

   This study aims to investigate the effect of visualization with neurofeedback on postoperative recovery in patients undergoing physical rehabilitation from 4 orthopedic surgical procedures: anterior cruciate ligament reconstruction (ACLR), total knee arthroplasty (TKA), total hip arthroplasty (THA), and hip arthroscopy (HA) for femoroacetabular impingement syndrome (FAIS). More specifically, neurofeedback training will be implemented using a novel technology developed by i-BrainTech™.

   The findings of this study have the potential to revolutionize physical rehabilitation protocols for patients, offering a novel approach that integrates visualization therapy with neurofeedback to enhance standard physical rehabilitation. This could lead to faster, more complete recoveries, and potentially mitigate the long-term impacts of AMI. The successful application of this technology would also help deepen current understanding of neuroplasticity, specifically the malleability of the neuromuscular pathways and how this can improve motor control.

   Purpose

   The purpose of this study is to investigate the effect of NFVT on postoperative recovery in patients rehabilitating from orthopedic surgeries.

   Hypothesis

   It was hypothesized that through targeted NFVT using i-BrainTech™, post-surgical participants will experience improved muscle activation, which in turn will contribute to better rehabilitation outcomes, strength, such as range of motion, and functional mobility. We also hypothesize that these improvements seen throughout the recovery period will have a positive impact on short-term patient-reported outcome surveys (PROs).
2. Methods

   Settings & Locations

   Conducted at Rush University Medical Center, specifically within:
   * The main campus of Midwest Orthopaedics at Rush (MOR) Sofija and Jorge O. Galante Orthopedic Building, 1611 W Harrison St, Chicago, IL 60612
   * Motion Laboratory in the MOR Orthopedic Building
   * Physical therapy facility (Chicago location)
3. Interventions

   Control group: Standard post-surgical rehabilitation therapy Intervention Group: Standard post-surgical rehabilitation therapy + i-BrainTech neurofeedback training
   * Procedure: Patients use EEG-based neurofeedback twice a week until 8 weeks post-operatively.
   * Neurofeedback setup: EEG cap monitors motor cortex activation, guiding visualization exercises
   * Training sessions: Patients visualize movements, and EEG feedback helps optimize motor activation

   Physical Therapy

   Patients will follow a standard physical therapy protocol. The protocol will be assigned by their respective surgeon who conducted the procedure and will be specific to the procedure that the patient underwent. The standardized physical therapy protocols will be attached in supplemental materials.

   Treatment Group Intervention:

   The main study intervention for the treatment group involves NFVT using the i-BrainTech™ Platform.

   This is a technology that uses electroencephalography (EEG) to read the electrical activities in the brain [7]. Active neurons in the brain causes change in electrical activities on the scalp, detectable by electrodes placed on the scalp. The sensing electrodes are completely passive, incapable of sending electrical current to the wearer. An EEG cap will be used with sensing electrodes aligned to the frontal cortex and the motor cortex. The detected electrical activity from these locations of the scalp will transmitted to the computer, which allows for assessment of focus and motor cortex activity [8]. There are multiple cap sizes to ensure a comfortable fit.

   By concentrating and imagining themselves performing the rehabilitation movements (visualization), patients activate their own motor and pre-frontal cortices. The EEG sensors detect the increased brain electrical activity, and the i-BrainTech™ software translates the EEG signal into a virtual avatar figure performing such movements on a computer monitor, providing feedback to the patients on their visualization efforts (neurofeedback). Patients will effectively play a video game using their own brain signals. By turning this feedback process into a video game, the i-BrainTech™ platform provides an incentive for the user to intensely focus and visualize the rehabilitation exercises, and in the process activate and strengthen the neural pathways responsible for these rehabilitation movements. The repeated activation of neural pathways theoretically improves their muscle control and reduces AMI [6].

   Instruction to Participants (how to play the "game")

   The i-BrainTech™ training station has a laptop and EEG caps. Participants will be seated in front of the laptop and put on the appropriately sized EEG cap. A conductive gel is injected into 2 insertion points on the cap. The column of gel touches the participant's skin on one side and the sensor on the other. The gel is water-soluble and dries up in chunks and is not sticky. The conductive gel is routinely used in the clinic and pre-operative area for ultrasound. The wet gel can be wiped off with a paper towel and the dried gel can be pulled off the participant's scalp as it does not stick to hair. The remaining fragments will be washed away when the patient showers.

   The session will be started and the i-BrainTech™ software will provide on screen prompts and feedback to the user.

   First is a 2-minute calibration period. During this time, the user is prompted to relax their mind so baseline brain activity may be detected. The brain activity above the baseline is used to control the cartoon avatar performing rehabilitation exercises.

   After calibration, a 20-minute NFVT session begins. Participants are prompted to imagine themselves performing various rehabilitation exercises (visualization). The selections of exercises are the rehabilitation exercises they will eventually perform at a physical therapy session, specific to their surgical procedures (Table 1). The software provides real time feedback on how concentrated the user is with the task, and how well the user is at visualizing the specific therapy exercises. The video game incentivizes participants to concentrate on the visualization therapy to maximize their score.

   When the participant finishes the i-BrainTech™ training session, they will remove the EEG cap and move on to their standard-of-care physical therapy session.
4. Clinic Flow and Timing of Assessments

   Participants in the intervention group will perform virtual rehabilitation exercises for 20 minutes 2 times per week for the first 8 weeks postoperatively.

   Approximately 45 minutes total is required for setup, calibration, virtual rehabilitation, and clean up.

   After the virtual rehab session, patients in the intervention group will move on to their standard-of-care PT session based on the surgeon's protocol specific to their operation. Patients in the control group go directly to their standard PT session.

   The intervention group will spend an additional 45 minutes in clinic to perform the i-BrainTech™ training session for a total study visit time of no more than 1-1.5 hours.

   The control group will spend 45 minutes to 1 hour of total study visit time.

   Participants will continue receiving their standard clinical care with their attending healthcare team throughout the study. In addition, they will attend scheduled study visits at the Motion Laboratory in the Orthopedic Building at Rush University Medical Center for motion analysis and physical testing at 2 months, 4 months, and 6 months post-surgery.

   At each visit, anthropometric data (age, height, and weight) will be collected first. Participants will then change into standardized clothing provided by the research team.

   Surface Electromyography (sEMG)

   sEMG data will be collected from five muscles: rectus femoris, vastus medialis oblique, vastus lateralis, semitendinosus, and biceps femoris, using a research-grade sEMG system. Electrode placement will follow the SENIAM (Surface EMG for a Non-Invasive Assessment of Muscles) protocol.

   Per SENIAM (www.seniam.org) guidelines, the skin will be shaved, lightly abraded with abrasion wipes, and cleaned with alcohol wipes before electrode application. Electrodes will be placed at least 2 cm apart to minimize crosstalk, and voluntary contractions will be performed to confirm correct placement.

   Each muscle will be assessed individually before data collection. Once all sensors are verified, simultaneous sEMG and 3D kinematic data collection will be performed using Qualisys Track Manager software or similar.

   Motion Capture

   To evaluate patient-specific movement mechanics, a markerless multi-camera motion analysis system will be used to track kinematics, while instrumented force plates will measure ground reaction forces. The markerless system allows for accurate motion tracking while significantly reducing setup time-by up to 80% since no physical markers need to be placed on the skin

   Participants will be evaluated while completing the following functional tasks.

   At 2 months postoperatively, all patients-regardless of the surgical procedure-will undergo motion analysis and strength testing. The motion analysis will include walking, bilateral squats, and a procedure-specific lunge (forward lunge for ACLR and TKA; lateral lunge for THA and hip arthroscopy). Strength assessments will focus on knee extension for ACLR and TKA, and hip extension and abduction for THA and hip arthroscopy.

   At 4 months postoperatively, all groups will repeat the same motion analysis tasks as at 2 months, with the addition of a single-leg vertical jump. Strength testing will now include two joint actions: knee extension and flexion for ACLR and TKA, and hip extension and abduction for THA and hip arthroscopy.

   At 9 months postoperatively, assessments will mirror those conducted at the 4-month follow-up for all surgical groups, including the same motion tasks and strength tests.

   This schedule allows for tracking recovery progression over time using both movement quality and strength performance.

   Strength testing

   Strength testing will be conducted after sEMG placement and motion analysis. Participants will keep the sEMG sensors on while performing maximum voluntary contractions (MVC) for knee flexion and extension.

   Isometric and isokinetic strength will be assessed using either a Biodex dynamometer or a handheld dynamometer, depending on equipment availability and participant-specific considerations. Strength data will also be used to normalize sEMG signals, with mean amplitudes of each phase expressed as a percentage of MVC. A 30% MVC normalization will be applied to allow for valid comparisons across groups.

   Total Testing Time

   The full testing session-including subject setup, EMG placement, motion analysis, and strength testing-will take approximately 30 to 45 minutes. Participants will be offered opportunities for water and seated rest breaks as needed throughout the session to ensure comfort and minimize fatigue.
5. Outcomes

   Primary outcomes

   ACLR and TKA
   * Outcome Measure Title

     o Knee extension strength
   * Outcome Measure Description
   * Maximal isokinetic knee extensor strength (Newtons/BMI). Maximal isokinetic knee extensor strength will be assessed using standardized dynamometry procedures with Biodex Isokinetic Dynamometer (Biodex System 3) at 2, 4 and 6 months after surgery. Each participant will perform three to five maximal voluntary isometric contractions of the knee extensors. The average of the peak torque values will be used for analysis. To account for individual differences in body size, values will be normalized to the participant's body mass index (Newtons/BMI). The first assessment will occur at 2 months to ensure patient safety and measurement consistency, as early postoperative conditions (e.g., pain, swelling) could compromise the reliability and validity of strength testing.
   * Outcome Measure Time Frame

     o 2, 4 and 6 months
   * Statistical Analysis

     * Linear mixed-effects models :
     * Linear mixed-effects models will be used to analyze changes in knee extensor strength between the intervention and control group across the 2-, 4-, and 6-month follow-up assessments. This approach accounts for repeated measures within participants and allows for the evaluation of group differences over time. Group (intervention vs. control), time (2, 4 and 6 months), and their interaction will be entered as fixed effects, with subject-level random intercepts. Significant main effects or interactions will be further examined using pairwise comparisons of estimated marginal means, with Tukey's adjustment for multiple comparisons to determine pairwise differences. All results will be reported with estimated means, p-values, and 95% confidence intervals. .

   Hip arthroscopy and THA
   * Outcome Measure Title

     o Hip Abduction Strength
   * Outcome Measure Description

     o Maximal isokinetic hip abductor strength (Newtons/BMI). Maximal isokinetic hip abductor strength will be assessed using standardized dynamometry procedures with Biodex Isokinetic Dynamometer (Biodex System 3) at 2, 4 and 6 months after surgery. Each participant will perform three to five maximal voluntary isometric contractions of the hip abductors. The average of the peak torque values will be used for analysis. To account for individual differences in body size, values will be normalized to the participant's body mass index (Newtons/BMI). The first assessment will occur at 2 months to ensure patient safety and measurement consistency, as early postoperative conditions (e.g., pain, swelling) could compromise the reliability and validity of strength testing..
   * Outcome Measure Time Frame

     o 2, 4 and 6 months
   * Statistical Analysis

     * Linear mixed-effects models :
     * Linear mixed-effects models will be used to analyze changes in hip abductor strength between the intervention and control group across the 2-, 4-, and 6-month follow-up assessments. This approach accounts for repeated measures within participants and allows for the evaluation of group differences over time. Group (intervention vs. control), time (2, 4 and 6 months), and their interaction will be entered as fixed effects, with subject-level random intercepts. Significant main effects or interactions will be further examined using pairwise comparisons of estimated marginal means, with Tukey's adjustment for multiple comparisons to determine pairwise differences. All results will be reported with estimated means, p-values, and 95% confidence intervals.

   Secondary outcomes are outlined in the supplementary material attached to this protocol and include EMG activation during functional tasks and strength tests; flexibility tests, PROs, and AMI classification
6. Statistical Methods

   Statistical methods are summarized in the supplementary material. For the primary outcome, linear mixed-effects models will be used to assess changes in knee and hip strength following ACLR, TKA, THA, and HA procedures. Strength outcomes will be compared between the intervention and control groups at 2, 4, and 6 months postoperatively. This modeling approach accounts for repeated measures within participants and allows for the evaluation of group differences over time. Group (intervention vs. control), time (2, 4 and 6 months), and their interaction will be entered as fixed effects, with subject-level random intercepts. Significant main effects or interactions will be further examined using pairwise comparisons of estimated marginal means, with Tukey's adjustment for multiple comparisons to determine pairwise differences. All results will be reported with estimated means, p-values, and 95% confidence intervals

   Secondary outcomes will follow a similar analytic approach using linear mixed-effects models, accounting for repeated measures and assessing group-by-time interactions, with appropriate post hoc testing as needed.

   To assess the time-series data of kinematics and kinetics across different conditions and time points, Statistical Parametric Mapping (SPM) will be utilized. SPM is a robust analytical approach that allows for the statistical evaluation of entire waveforms, reducing the limitations of discrete-point analysis in biomechanical research. SPM maintains the temporal structure of the data and enables the identification of significant differences across the entire movement cycle, offering a more comprehensive understanding of biomechanical adaptations post-surgery.

   SPM will be applied to joint angle waveforms, ground reaction forces, and external moment profiles to compare surgical groups, timepoints, and control conditions. This approach will help detect subtle but functionally relevant alterations in movement patterns that may not be captured using traditional peak or mean value analyses.

   Kinematic and kinetic data will be collected bilaterally to examine compensatory strategies in the contralateral limb. EMG and strength only in the affect side. The integration of markerless motion capture, inverse dynamics, and SPM analysis will provide a detailed and objective assessment of post-surgical movement patterns.

   Differences in the distribution of knee AMI classification (grades 0-3) between groups will be assessed using Fisher's exact test.

   Statistical significance for all analyses will be set at an a priori α of 0.05. All data analyses will be completed using R version 4.2.3 (R Core Team).

   Loss to Follow Up

   Data analysis will be conducted according to the intention-to-treat (ITT) principle. Patients who are lost to follow-up for any reason will be included in the primary analysis using the last observation carried forward (LOCF) method.
7. Power Analysis

   Strength

   Separate power analyses were conducted for the knee surgery cohort (ACL and TKA) and the hip surgery cohort (HA and THA).

   Knee Surgery (ACL and TKA)

   The power analysis for the knee surgery group was based on data from a previous randomized controlled trial, which evaluated the effects of motor imagery on quadriceps strength following total knee arthroplasty (TKA). The original study included 12 patients with unilateral TKA, assessed six months postoperatively (10 females, 2 males). The primary outcome was quadriceps maximum voluntary isometric contraction (MVIC), measured using a hand-held dynamometer. This method is highly correlated with the Biodex system currently used in the present trial (R = 0.91).

   Statistical analysis was performed in R version 4.3.2 using the pwr package. The mean quadriceps MVIC reported was 20.58 N/BMI (SD = 1.85). Assuming a two-group parallel design (intervention vs. control) with 30 participants per group (total n = 60), the study is powered at 80% to detect a between-group difference of 1.31 N/BMI at a two-tailed α = 0.05 (adjusted α = 0.025 to account for multiple comparisons). This corresponds to a minimum detectable difference (MDD) of 6.31% between groups.

   Hip Surgery (HA and THA)

   The power analysis for the hip surgery group was based on data from a retrospective study, which evaluated hip abductor strength before and three months after hip arthroscopy for femoroacetabular impingement (FAI). The study included 29 individuals (mean age 27.4 ± 7.5 years; 76% female). The primary outcome was hip abductor MVIC, also measured with a hand-held dynamometer.

   The reported mean abductor MVIC was 1.97 N/kg (SD = 0.42). A two-group parallel design with 30 participants per group (n = 60 total) provides 80% power to detect a between-group difference of 0.31 N/kg at a two-tailed α = 0.05 (adjusted α = 0.025). This represents an MDD of 15.6%.

   To contextualize the clinical relevance of the estimated minimal detectable differences (MDDs), previously published values for minimal clinically important differences (MCIDs) were reviewed. For quadriceps MVIC, a previous study reported an MCID of 26.9% in older adults with COPD, with improvements associated with enhanced performance in the six-minute walk test. In patients undergoing ACL reconstruction, a limb strength asymmetry of 10% is considered a clinically relevant threshold and a predictor of reinjury. For hip abductor strength, although there is no universally accepted MCID after hip surgery, many studies consider a relative difference of 10-15% to be clinically meaningful. These values serve as important clinical benchmarks and support the interpretation that the proposed sample size (n = 60 per pathology group) is adequate to detect both statistically and clinically relevant between-group differences in strength outcomes.

   Kinematics

   A separate power analysis was conducted for the secondary kinematic outcomes to estimate the minimum detectable differences achievable with the current sample size and 80% statistical power. This analysis helps ensure that the study is adequately powered to detect changes that are not only statistically significant but also clinically meaningful.

   The power analysis was based on data from a previous investigation conducted in the same laboratory where the current study will take place, using identical equipment, camera setup, and software configuration parameters. Individuals assessed in study were 5 healthy males (mean age 26) and 5 females (mean age 28) (n=10). The primary variables of interest for the power analysis were the knee peak flexion angle (for the ACL and TKA study arms) and the hip peak extension angle (for the hip arthroscopy and THA study arms) during the gait cycle, measured using a markerless motion capture system (Theia 3D, Theia Markerless Inc., Kingston, ON). The statistical analysis was conducted using R version 4.3.2 (R Core Team, 2023) and the pwr package (Champely, 2020).

   For the knee flexion angle, a previous investigation reported a mean of 19° with a standard deviation (SD) of 7.68°. Using these values, a two-group parallel design with 30 participants per group (total n = 60) was powered at 80% to detect a between-group difference of at least 5.65° at a two-sided α = 0.05 (adjusted α = 0.025 for sidedness). Similarly, for hip extension angle (mean = 9.25°, SD = 5.11°), the same sample size and power would yield a minimum detectable difference of 3.76°.

   To contextualize the clinical relevance of the estimated minimal detectable differences (MDDs), previously published values for minimal clinically important differences (MCIDs) were reviewed. For knee flexion angle, a previous study reported an MCID of 6.81 degrees based on gait analysis of the unaffected limb in stroke patients. In a different clinical context, another study identified an MCID of 5 degrees for passive range of motion following total knee arthroplasty, with improvements in flexion associated with better knee function and higher patient satisfaction. Regarding hip extension angle, it was established an MCID of 2.86 degrees in stroke patients using motion analysis of the unaffected limb. These values serve as clinical benchmarks to interpret the statistical power and meaningfulness of the differences targeted in this study.
8. Randomization

   Sequence Generation

   Randomized list generation before trial commencement utilizing the National Institute of Health (NIH) Clinical Trial Randomization Tool. A 1:1 allocation (intervention vs. Control) per procedure will be implemented.

   The randomization sequence will be generated before trial commencement by an independent data manager using the Clinical Trial Randomization Tool developed by the National Cancer Institute (NCI). The tool will use the Asymptotic Maximal procedure, a restricted randomization method that limits the imbalance between trial arms to a pre-specified Maximum Tolerated Imbalance (MTI) of 3. The randomization list will be created for a total of 70 participants, with no stratification applied.

   Type of Randomization

   A simple two-arm parallel group design will be used with a 1:1 allocation ratio for each procedure (ACLR, THA, TKA, and HA), with a separate randomization list of 35 participants per group (total n=70) generated independently for each procedure. Each procedure will be treated as a distinct trial with its own allocation sequence. The final participants will be randomly assigned in accordance with the MTI threshold, allowing minor tolerable imbalances between arms. No stratification or blocking will be implemented. The increased sample size per group (n=35 instead of n=30) accounts for potential losses or allocation issues during the study. Additional allocation slots beyond the target sample size will be generated to account for unexpected exclusions, dropouts before randomization, or technical errors during allocation.

   Allocation Concealment Mechanism

   Allocation concealment will be ensured using the REDCap (Research Electronic Data Capture) Randomization Module, which provides a secure, centralized, and automated platform for treatment allocation. The randomization sequence will be generated and implemented within REDCap by an independent data manager who will not be involved in participant enrollment, intervention, and outcome assessment. The system will be configured to assign participants in real time only after eligibility has been confirmed and baseline data have been entered, thereby preventing any foreknowledge of the upcoming assignment. Investigators, study staff, and participants will remain unaware of the allocation sequence prior to assignment. REDCap's access controls and audit logs will safeguard against manipulation and preserve allocation concealment throughout the trial.

   Implementation

   All patients referred for ACLR, TKA, THA, or HA procedures in the physician's office will be referred to the research team to assess eligibility criteria and initiate the enrollment process, either in person or by phone. Eligible patients will be enrolled in the study during the pre-operative period and will complete baseline assessments. Following surgery, participants will be assigned to one of the intervention groups one day prior to the intervention date. Group allocation will be performed by an independent data manager using the REDCap Randomization Module and communicated only to the team responsible for delivering the NFVT. The individual responsible for generating the allocation sequence will be distinct from those involved in enrolling participants and assigning interventions.

   Blinding

   Investigators and physicians will be blinded to group allocation to minimize bias in clinical decision-making and post-operative care. Patients will not be blinded due to the nature of the neurofeedback intervention, which cannot be masked. Both study groups will receive standard rehabilitation, with the only difference being the addition of NFVT in the intervention arm. The neurofeedback sessions will take place within the physical therapy clinic, immediately prior to scheduled physical therapy appointments.

   The team delivering the neurofeedback intervention will be the only personnel aware of group allocation. Treating physicians, physical therapists, outcome assessors, and the statistical analysis team will remain blinded to participant allocation throughout the trial. Statistical analyses will be performed by the Rush Statistical Analysis team, an independent third-party ancillary resource, using a coded dataset to ensure blinding is maintained during data analysis.

   Unblinding Procedures

   Given the non-invasive nature of the EEG-based neurofeedback intervention, adverse effects are not expected. However, in rare cases where unblinding is required-such as equipment malfunction, unexpected clinical events, or participant withdrawal-a formal request must be submitted to the principal investigator (PI) or Data and Safety Monitoring Board (DSMB). All unblinding events will be logged with justification and date.

   For emergencies, a dedicated study coordinator will have secure access to the REDCap randomization module and group allocation. This coordinator will be available to authorized clinical staff in urgent scenarios requiring immediate unblinding. Outcome assessors and data analysts will remain blinded throughout the study.

   These procedures align with CONSORT guidelines and will be included in staff training to ensure adherence.
9. Recruitment

The investigators will identify eligible patients in the clinic, and the research study staff will discuss the study with eligible patients. The informed consent process may occur over a period of several discussions, culminating in the signing of a consent form in the office (iPad) or sent to their verified email address.

Informed consent will be obtained via the eConsent process through the secured platform Patient IQ. The patient will be prompted to reply with the appropriate passcode to access the consent form and then provide the passcode again with their signature (secured). A copy of the time stamped document will be sent to the study team through the electronic platform and a copy will be sent to the participant. All participants will be consented prior to surgery and the performance of research related testing activities.

ELIGIBILITY:
Participants

* Inclusion Criteria:

  * Patient age >18 years
  * Ability to complete neurofeedback training and follow study follow-ups
  * Indicated for one of the four investigated orthopedic procedures
* Exclusion Criteria:

  * Inability to participate in neurofeedback training
  * Lack of decisional capability
  * History of stroke, movement disorder (e.g. Parkinson's), peripheral neuropathy
  * Cardiac pacemaker or other internal electronic device
  * BMI >35
  * Previous surgery or specific pathology on the affected joint (refer to procedure specific indications below)

Procedure Specifics:

Anterior cruciate ligament reconstruction (ACLR) Procedure-specific Inclusion Criteria

* Patients undergoing primary ACLR with autograft or allograft tissue
* Adjunct lateral Extra-articular tenodesis will be included
* Additional meniscus debridement and repair will be included Procedure-specific exclusion criteria
* Revision ACL surgery
* Moderate to Severe arthritis - Kellgren-Lawerence (KL) Grade > 3
* Patients with meniscus root repair
* Non-weight-bearing status exceeding 1 week postoperatively

Total knee arthroplasty (TKA) Procedure specific inclusion criteria

* Patients undergoing primary TKA
* Preoperative total knee range of motion of at least 100 degrees (combined flexion and extension)
* Prior extensor mechanism tendon repair, quadriceps or patella tendon. Procedure specific exclusion criteria
* Revision surgery
* Hinged implant
* Any open procedure involving the knee joint
* Symptomatic arthritis in the contralateral knee with planned or expected total knee arthroplasty within 6 months
* Inflammatory Arthritis

Total hip arthroplasty (THA) Procedure Specific Inclusion Criteria

* Patients undergoing primary THA Procedure Specific Exclusion Criteria
* Revision Surgery
* Any open procedure involving the hip joint
* Bilateral THA procedures
* Inflammatory Arthritis

Hip arthroscopy (HA) for femoroacetabular impingement syndrome (FAIS) Procedure Specific Inclusion Criteria

· Patients undergoing HA for FAIS Procedure Specific Exclusion Criteria

* Revision Surgery
* Diagnosis of hip dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Knee extensor strength | 2, 4 and 6 months
  ACLR and TKA groups: Maximal isokinetic knee extensor strength (Newtons/BMI). Maximal isokinetic knee extensor strength will be assessed using standardized dynamometry procedures with Biodex Isokinetic Dynamometer (Biodex System 3) at 2, 4 and 6 months after surgery. Each participant will perform three to five maximal voluntary isometric contractions of the knee extensors. The average of the peak torque values will be used for analysis. To account for individual differences in body size, values will be normalized to the participant's body mass index (Newtons/BMI). Body Mass Index (BMI) = weight (kg) / [height (m)]². The first assessment will occur at 2 months to ensure patient safety and measurement consistency, as early postoperative conditions (e.g., pain, swelling) could compromise the reliability and validity of strength testing.
Hip Abductor Strength | 2, 4 and 6 months
  Hip arthroscopy and THA: Maximal isokinetic hip abductor strength (Newtons/BMI). Maximal isokinetic hip abductor strength will be assessed using standardized dynamometry procedures with Biodex Isokinetic Dynamometer (Biodex System 3) at 2, 4 and 6 months after surgery. Each participant will perform three to five maximal voluntary isometric contractions of the hip abductors. The average of the peak torque values will be used for analysis. To account for individual differences in body size, values will be normalized to the participant's body mass index (Newtons/BMI). Body Mass Index (BMI) = weight (kg) / [height (m)]². The first assessment will occur at 2 months to ensure patient safety and measurement consistency, as early postoperative conditions (e.g., pain, swelling) could compromise the reliability and validity of strength testing.

SECONDARY OUTCOMES:
Joint Kinematics During Functional Tasks (Walk, Lunge, Bilateral Squats, Single Leg Vertical Jump) | 2, 4 and 6 months
  Hip, knee, ankle, trunk, pelvis, thigh, shank, trunk, and foot angles during walk, lunge, bilateral squats, and single-leg vertical jump.
  Reported as continuous waveforms over the task cycle (angles vs. % of task cycle).
Joint Kinetics During Functional Tasks (Walk, Lunge, Bilateral Squats, Single Leg Vertical Jump) | 2, 4 and 6 months
  External and internal moments at the hip, knee, and ankle in the sagittal, frontal, and transverse planes.
  Unit of Measure: Joint moment expressed as a percentage of body weight times height (%BW·HT). Reported as continuous waveforms over the task cycle (%BW·HT vs. % of task cycle).
EMG Amplitude of Lower Limb Muscles During Functional Tasks | 2, 4 and 6 months
  Normalized EMG amplitude (mean and maximum) of the vastus lateralis, rectus femoris, vastus medialis, semimembranosus, semitendinosus, gluteus maximus and gluteus medius during walking, squats, lunge, single-leg vertical jump and strength tests.
  Unit of Measure: % Maximum Voluntary Contraction (%MVC)
Flexibility | 2, 4 and 6 months
  TKA and ACLR:
  Passive knee flexion range of motion Passive knee extension range of motion
  THA and HA:
  Thomas test Passive internal/external rotation range of motion
  Unit of measure: degrees
International Knee Documentation Committee (IKDC) Subjective Knee Form | Pre-operative, 2, 4 and 6 months, 1 year, 2 years
  ACLR group:
  Description: A knee-specific outcome measure assessing symptoms, function, and sports activity. Scores range from 0 to 100; higher scores indicate better knee function.
  Unit of Measure: Units on a scale (0-100)
Knee and Hip Strength | 2, 4 and 6 months
  Maximum torque generated during isokinetic and isometric hip extension and knee flexion, reported as raw and BMI-normalized values.
  Unit of Measure: Newton-meters (Nm); Nm/kg/m²
Area Under the Curve of Muscle Activation During Functional Tasks | 2, 4, and 6 months
  Area under the EMG curve (AUC) for each muscle during walking, squats, lunge, and single-leg vertical jump, representing total activation over the task. Unit of Measure: %MVC × seconds
Torque Curves of Hip and Knee During Flexion, Extension, Abduction | 2, 4 and 6 months
  Full torque trace over the range of motion during contractions of hip and knee. Unit of Measure: Newton-meters across % range of motion
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR and TKA Groups:
  Description: Short-form knee-specific outcome measure evaluating stiffness, pain, and physical function. Scores range from 0 to 100; higher scores indicate better function.
  Unit of Measure: Units on a scale (0-100)
Veterans RAND 12-Item Health Survey (VR-12) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR, TKA, and THA groups:
  Description: General health survey assessing physical and mental health components. Norm-based scoring with mean = 50 and SD = 10; higher scores indicate better health.
  Unit of Measure: Units on a scale (norm-based)
Patient-Reported Outcome Measurement Information System - Pain Interference (PROMIS-PI) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR and HA groups:
  Description: Assesses how pain interferes with daily activities. T-scores range from 0 to 100; higher scores indicate greater pain interference.
  Unit of Measure: T-score (0-100)
Patient-Reported Outcome Measurement Information System - Physical Function (PROMIS-PF) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR and HA groups:
  Description: Assesses physical function ability in daily life. T-scores range from 0 to 100; higher scores indicate better function.
  Unit of Measure: T-score (0-100)
PROMIS Depression Short Form | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR and HA groups:
  Description: Evaluates symptoms of depression. T-scores range from 0 to 100; higher scores indicate more severe depressive symptoms.
  Unit of Measure: T-score (0-100)
Anterior Cruciate Ligament - Return to Sport after Injury Scale (ACL-RSI) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR group:
  Description: Assesses psychological readiness to return to sport after ACL injury. Scores range from 0 to 100; higher scores indicate greater readiness.
  Unit of Measure: Units on a scale (0-100)
Tampa Scale for Kinesiophobia - 11-item Version (TSK-11) | Time Frame: Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACRL, THA, TKA and HA groups. Description: Measures fear of movement/re-injury. Scores range from 11 to 44; higher scores indicate greater fear of movement.
  Unit of Measure: Units on a scale (11-44)
Knee Society Score (KSS) | Time Frame: Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  TKA group. Description: Clinician- and patient-reported outcome assessing pain, function, range of motion, and stability after total knee arthroplasty. Scores range from 0 to 100; higher scores indicate better outcomes.
  Unit of Measure: Units on a scale (0-100)
Knee Single Assessment Numeric Evaluation (Knee SANE Score) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  ACLR group:
  Description: Single-question assessment where patients rate their knee function as a percentage of normal (0-100%). Higher scores indicate better function.
  Unit of Measure: Percentage (0-100%)
Forgotten Joint Score-12 (FJS-12) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  TKA and THA groups: Description: Patient-reported measure of joint awareness in daily life. Scores range from 0 to 100; higher scores indicate less awareness of the artificial joint and better outcome.
  Unit of Measure: Units on a scale (0-100)
EuroQol 5-Dimension 3-Level Questionnaire (EQ-5D-3L) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  TKA and THA groups:
  Description: Generic measure of health-related quality of life across five domains. Reported as an index score (range: -0.594 to 1) and/or visual analog scale (VAS; 0-100). Higher scores indicate better health status.
  Unit of Measure: Utility score (-0.594 to 1) and/or VAS (0-100)
Hip Dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS Jr) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  THA group:
  Description: Short-form patient-reported measure evaluating hip pain and physical function in patients undergoing joint replacement. Scores range from 0 to 100; higher scores indicate better hip function.
  Unit of Measure: Units on a scale (0-100)
Harris Hip Score (HHS) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  THA group:
  Description: Clinician-administered measure evaluating pain, function, deformity, and range of motion of the hip. Scores range from 0 to 100; higher scores indicate better hip function.
  Unit of Measure: Units on a scale (0-100)
12-item International Hip Outcome Tool (iHOT-12) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  Hip Arthroscopy (HA) group:
  Description: Patient-reported measure assessing health-related quality of life in young, active patients with hip disorders. Scores range from 0 to 100; higher scores indicate better quality of life.
  Unit of Measure: Units on a scale (0-100)
Hip Outcome Score (HOS) | Pre-operative, 2, 4, and 6 months; 1 year; 2 years
  HA group:
  Description: Patient-reported outcome evaluating hip function, combining items related to daily and sports activities into an overall composite score. Scores range from 0 to 100; higher scores indicate better overall hip function.
  Unit of Measure: Units on a scale (0-100)

OTHER OUTCOMES:
Knee AMI Classification | 2, 4 and 6 months
  Sonnery-Cottet et al. knee AMI classification (Grade 0-3)
Digital Avatar Performance Metrics | 0 to 8 weeks of training
  Performance metrics generated during the neurofeedback training sessions will be collected directly from the iBrainTech software. Attention, motor imagery, and session scores.
Spatiotemporal Gait Parameters | 2, 4, and 6 months
  Stride length, step length, cadence, gait speed, stance time, swing time, and double support time during walking task.
EMG Timing of Muscle Onset and Offset During Functional Tasks | 2, 4 and 6 months
  Onset and offset timing of activation of key muscle groups during walking, squats, lunge, and single-leg vertical jump. Unit of Measure: % of task cycle
Co-Contraction Index Between Quadriceps and Hamstrings During Functional Tasks | 2, 4, and 6 months
  Quadriceps-to-hamstrings co-contraction index calculated during walking, squats, lunge, and single-leg vertical jump. Unit of Measure: Unitless index value

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Chahla, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT07020312/Prot_SAP_000.pdf